CLINICAL TRIAL: NCT04568057
Title: Effect of Transcranial Near Infrared Light 1068 nm Upon Memory Performance in Ageing Healthy Individuals: a Pilot Study.
Brief Title: Effect of Transcranial NIR Light Upon Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maculume Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M20Q004
Record Dates: First submitted 2020-09-22; First posted 2020-09-29 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2020-09

CONDITIONS: Age-related Cognitive Decline
Keywords: ageing; photobiomodulation; transcranial

STUDY DESIGN:
Intervention Model Description: Double-blind placebo-controlled, one group received a placebo device and once group an active device.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: NIR light is invisible to the human eye, therefore the placebo units will operate in an identical manner to that of the active units.
  The active and placebo helmets will look identical and their external operation will appear identical, each device will be marked with a code by the manufacturer, there will be no way to identify a device from active or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIR Transcranial phototherapy device (Active Comparator): The active transcranial phototherapy device. 1068 nm NIR Transcranial phototherapy PBM-T device An air-cooled LED helmet with a peak wavelength of 1068 nm, spectral width of 60 nm, and a 6-minute internal timer was used. The average optical power output of the combined arrays is circa 3.8 Watts, 12mw/sq. cm. The total energy to be delivered to the cranium is 1368J (3.8 x 360) per treatment session.
  Interventions: Device: NIR Transcranial phototherapy device
- Placebo Device. (Placebo Comparator): Placebo cranial device. The external appearance of the device is identical to that of the active device but no NIR light is emitted.
  Interventions: Device: Placebo Transcranial Device

INTERVENTIONS:
Device: NIR Transcranial phototherapy device — 1068 nm NIR helmet
  Arms: NIR Transcranial phototherapy device
Device: Placebo Transcranial Device — The placebo device looks like the active device.
  Arms: Placebo Device.

SUMMARY:
A double-blind placebo-controlled study evaluating the effect of 1068nm NIR trans-cranial phototherapy upon the cognitive function of healthy individuals between the age of 45 years and 80 years.

DETAILED DESCRIPTION:
Interested participants will be sent a participant information bundle consisting of the participant information sheet, consent document, and data collection sheets. One week after receiving these documents, they will be contacted by a member of the research team to ascertain if they wish to participate. If the individual wishes to participate in the trial, an appointment at a mutually convenient time will be made for the volunteer to be seen. The initial screening interview will be conducted by a trained research assistant. At this appointment, the research assistant will explain the details of the trial and offer an opportunity for the volunteer to ask questions. The consent document will then be completed by the volunteer and countersigned by the researcher.

1. The volunteer will have several days to decide whether they wish to participate in the trial as they will have received the information pack in the mail previously. The volunteer would have the option of speaking to the Investigator directly before enrolling.
2. The volunteer will have an opportunity to ask questions and have any points of concern clarified.
3. Informed consent will be obtained from the volunteer.
4. The volunteer will be interviewed and a detailed history is taken. Baseline information regarding the volunteer's circumstance will be gathered, including confirming the MMSE score is >28 (a score of <28 is an exclusion criterion).
5. The volunteer will be allocated a number and will we offered a choice of appointment times and will be seen on three separate occasions for assessment of their executive function and memory. Three tests are necessary to average the day-to-day variation present in cognitive functioning.
6. Testing will be rescheduled if the volunteer has a minor intercurrent illness eg. Flu, minor viral infection.
7. After the third ANAM assessment the volunteer will proceed to receive the intervention.
8. Intervention procedure: Once allocated to either active or placebo group everyone will be given a trans-cranial intervention device to take home with them. They will be shown how to use the device, which should be used for 6 minutes twice daily every day of the week.
9. Telephone contact will be made by a researcher with the participant every 2 weeks throughout the intervention period to make the following verbal observations:

a. has there been any change in the health of the participant? b. Are there any problems with the device? j. After 56 days of twice-daily intervention, the participant will be scheduled for re-assessment on three separate days. They will continue with the use of the NIR helmet device until the last assessment is completed.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥45 years, ≤ 80 years
* MMSE score >28 (out of 30)
* No chronic illnesses other than hypertension, asthma, or mild COPD
* Stable, controlled chronic illness e.g. hypertension, asthma, COPD

Exclusion Criteria:

* Diagnosed actively growing intracranial pathology (tumors etc.)
* Mental health illness
* Misuse of illegal substances or alcohol
* Use of regular systemic steroids or cancer drugs
* Cancers that affect your body
* Not fluent in English
* Depressed, or feeling depressed.
* Epilepsy
* Lacking capacity to give informed consent
* Previous history of stroke
* History of aggression or violence
* Inability to attend the research venue for assessment
* Assessed as probably being non-complaint with the intervention regime
* Diabetes
* Diagnosed with a neurological condition eg. Parkinson's disease, multiple sclerosis
* Diagnosed with dementia of any cause
* Chronic pain disorders
* Volunteers taking medication which would impair cognitive function such as gabapentin, pregabalin, strong opiates (e.g. morphine)
* Any chronic illness other than hypertension, asthma, or mild COPD.
* Not being available for all the assessment sessions.
* Participants currently involved in any other research program

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Automated Neuropsychological Assessment Metrics | 56 days
  Computerised neurophysiological assessment tool

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Dougal, MB ChB, Principal Investigator — Maculume Ltd.
Locations (1):
- Maculume Ltd, Spennymoor, Durham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hawkins KA, Jennings D, Vincent AS, Gilliland K, West A, Marek K. Traditional neuropsychological correlates and reliability of the automated neuropsychological assessment metrics-4 battery for Parkinson's disease. Parkinsonism Relat Disord. 2012 Aug;18(7):864-70. doi: 10.1016/j.parkreldis.2012.04.021. Epub 2012 May 18. PMID 22609082
- [Background] Jones WP, Loe SA, Krach SK, Rager RY, Jones HM. Automated neuropsychological assessment metrics (ANAM) and Woodcock-Johnson III Tests of Cognitive Ability: a concurrent validity study. Clin Neuropsychol. 2008 Mar;22(2):305-20. doi: 10.1080/13854040701281483. PMID 17853133
- [Background] Naeser MA, Zafonte R, Krengel MH, Martin PI, Frazier J, Hamblin MR, Knight JA, Meehan WP 3rd, Baker EH. Significant improvements in cognitive performance post-transcranial, red/near-infrared light-emitting diode treatments in chronic, mild traumatic brain injury: open-protocol study. J Neurotrauma. 2014 Jun 1;31(11):1008-17. doi: 10.1089/neu.2013.3244. Epub 2014 May 8. PMID 24568233
- [Background] Barrett DW, Gonzalez-Lima F. Transcranial infrared laser stimulation produces beneficial cognitive and emotional effects in humans. Neuroscience. 2013 Jan 29;230:13-23. doi: 10.1016/j.neuroscience.2012.11.016. Epub 2012 Nov 27. PMID 23200785
- [Derived] Dougal G, Ennaceur A, Chazot PL. Effect of Transcranial Near-Infrared Light 1068 nm Upon Memory Performance in Aging Healthy Individuals: A Pilot Study. Photobiomodul Photomed Laser Surg. 2021 Oct;39(10):654-660. doi: 10.1089/photob.2020.4956. PMID 34662523